CLINICAL TRIAL: NCT02130479
Title: Testing a Promising Treatment for Youth Substance Abuse in a Community Setting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA034064-01A1 (NIH)
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Substance Abuse; Delinquency; Mental Health
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management-Family Engagement (Experimental): The Contingency Management-Family Engagement or CM-FAM model integrates behavioral (e.g., drug testing linked with consequences) and cognitive behavioral (e.g., functional analyses of drug use, self-management and drug refusal skills training) strategies based on the Community Reinforcement Approach with effective family engagement strategies used in Multisystemic Therapy.
  Interventions: Behavioral: Contingency Management-Family Engagement
- Treatment as Usual (Active Comparator): Standard community-based substance abuse treatment services.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Contingency Management-Family Engagement
  Arms: Contingency Management-Family Engagement
Behavioral: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
This study aims to address a serious public health problem (i.e., substance abusing adolescents) by testing the effectiveness of a promising substance abuse treatment implemented in a community-based treatment setting (CM-FAM, a family-based contingency management intervention) in comparison to usual treatment services.

DETAILED DESCRIPTION:
The overriding purpose of the randomized trial is to examine the effectiveness of a promising and efficient outpatient treatment of adolescent substance abuse delivered in a community-based treatment setting. Although several evidence-based treatments of adolescent substance abuse are emerging, none have experienced widespread adoption in community settings. Thus, as noted by the Institute of Medicine (1998) more than a decade ago and reiterated more recently, a considerable science-service gap exists in regards to treatment of substance abuse in adolescents and adults.

For the proposed study, 204 adolescents meeting diagnostic criteria for substance abuse or dependence will be randomized to either the Contingency Management-Family Engagement (CM-FAM) or Treatment as Usual (TAU) conditions. A multimethod, multirespondent approach will be used to track clinical outcomes at 3, 6, 9, 12, and 18 months post recruitment. Clinical level outcomes pertain to youth substance use, criminal behavior, mental health functioning, and key mediators of serious antisocial behavior in adolescents (e.g., self-control, parental supervision, association with deviant peers). In addition, the incremental cost of CM-FAM will be determined for use in cost effectiveness analyses.

Aim 1: Over an 18-month post-recruitment follow-up, determine the relative effectiveness of CM-FAM vs. TAU in reducing adolescent participants' substance use, criminal activity (including incarceration), and mental health symptoms; and evaluate the cost effectiveness of CM-FAM in achieving these outcomes.

Aim 2: Examine possible moderators and mediators of intervention effectiveness. Moderator variables will include youth demographic and clinical (e.g., co-occurring disorders) characteristics. Mediator variables will include measures of self-control, parenting, and association with deviant peers - constructs targeted by CM-FAM.

ELIGIBILITY:
Inclusion Criteria:

* Age of 12-17 years
* Meeting criteria for substance use or abuse.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in youths' substance abuse frequency as measured by Urine Drug Screens and the Global Appraisal of Individual Needs Scale | Youth baseline, 3, 6, 9, 12, & 18 months post-baseline
Change in youths' delinquent behavior as measured by Juvenile Justice Archival Records and the Self-Report Delinquency Scale | Youth baseline, 3, 6, 9, 12, & 18 months post-baseline
Change in youths' mental health functioning as measured by the Brief Problem Checklist | Youth baseline, 3, 6, 9, 12, & 18 months post-baseline

SECONDARY OUTCOMES:
Change in youths' peer relations as measured by the Peer Delinquency and Drug Activities Scales, the Conventional Activities of Peers Scale, and the Bad Friends Scale from the Pittsburgh Youth Study | Youth baseline, 3, 6, 9, 12, & 18 months post-baseline
Change in family functioning as measured by the Caregiver Supervision Scale, the Discipline Scale, and the Communication Form from the Pittsburgh Youth Study | Youth baseline, 3, 6, 9, 12, & 18 months post-baseline
Change in youths' self-control as measured by the Good Behavioral Self-Control and the Poor Behavioral Regulation Scales | Youth baseline, 3, 6, 9, 12, & 18 months post-baseline

OTHER OUTCOMES:
Incremental costs associated with CM-FAM as measured by the Drug Abuse Treatment Cost Analysis Program | 6, 18, and 30 months following initiation of CM-FAM delivery
Change in youths' treatment duration and rates of completion as measured by clinic records | 6, 18, and 30 months following initiation of CM-FAM delivery
Change in therapists' perceptions of the functioning of their treatment facility as measured by the Organizational Readiness for Change Scale | Therapist baseline, 6, 12, 18, 24, & 30 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Scott Henggeler, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Circle Park Behavioral Health Services, Florence, South Carolina, United States